CLINICAL TRIAL: NCT07257107
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation Combined With Upper Extremity Robot-Assisted Training on Upper Extremity Motor Functions in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, rustem mustafaoglu, associate professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1277364
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Stroke Treatment; Stroke
Keywords: Stroke; Upper Extremity Robot-Assisted Training; Transcutaneous Auricular Vagus Nerve Stimulation; taVNS
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotics Assisted Education + taVNS (Active Comparator)
  Interventions: Device: Robotics Assisted Education + taVNS
- Robotics Assisted Education + sham (Sham Comparator)
  Interventions: Other: Robotics Assisted Education + sham

INTERVENTIONS:
Device: Robotics Assisted Education + taVNS — Conventional rehabilitation will be administered 3 days a week, 45 minutes per day, for 5 weeks. The combination of Upper Extremity Robotic-Assisted Training and Transcutaneous Auricular Vagus Nerve Stimulation will be administered 2 days a week, 45 minutes per day, for 5 weeks.
  Arms: Robotics Assisted Education + taVNS
Other: Robotics Assisted Education + sham — Conventional rehabilitation will be administered 3 days a week, 45 minutes per day, for 5 weeks. The combination of Upper Extremity Robotic-Assisted Training and Sham Transcutaneous Auricular Vagus Nerve Stimulation will be administered 2 days a week, 45 minutes per day, for 5 weeks.
  Arms: Robotics Assisted Education + sham

SUMMARY:
The effects of stroke on the upper extremity are a common and significant cause of long-term disability, with 65% of patients reporting an inability to participate in daily activities with the affected upper extremity after 6 months. Robotic-assisted training (RAT) has been widely used in recent years to improve upper extremity function. RAT positively impacts upper extremity function and activities of daily living by inducing motor learning from intense, highly repetitive, and task-focused movements of the upper extremity. However, current, limited clinical solutions, including minimally invasive transcutaneous auricular vagus nerve stimulation (taVNS), have not yielded promising results. Therefore, the aim of this study was to investigate the effects of the combination of taVNS and RTA on motor impairment, upper extremity motor function, grip strength, daily living characteristics, and quality of life in individuals with stroke. Stroke medications were randomly assigned to RDE+taVNS (n=15) and RDE+sham taVNS (n=15). All participants will receive conventional treatment for 45 minutes per day, 3 days per week, for 5 weeks. One group will also receive RDE+taVNS treatment for 45 minutes per day, 2 days per week, for 5 weeks, while the other group will receive RDE+sha taVNS. Participants will be assessed using the Fugl-Meyer Upper Extremity Assessment, ARAT (Action Research Arm Test), and Box and Block Test as primary outcomes at baseline and after 5 weeks.

This project will contribute to the literature by demonstrating the effectiveness of taVNS, one of the most promising methods available. Furthermore, the results will prompt discussion on the applicability of the method not only to stroke patients but also to other disease groups. The unique value of this project is that it is the first study to investigate product improvements in taVNS systems.

ELIGIBILITY:
Inclusion Criteria:

* 1) Individuals aged 18-70 years diagnosed with ischemic or hemorrhagic stroke lasting longer than 6 months,
* Moderate to severe upper extremity weakness (20-50 out of 66 on the Fugl-Meyer Upper Extremity Motor Assessment Scale),
* Ability to communicate and understand (Mini Mental State Examination (MMSE) score ≥ 23), and 4) Upper extremity spasticity of 2 or less on the Modified Ashworth Scale.

Exclusion Criteria:

* Use of any stimulation device, such as a pacemaker or other neurostimulator,
* Presence of a medical or cognitive condition (personality disorder, anxiety, depression, etc.) that would prevent participants from participating in the study,
* Receiving a Botox injection into the affected upper extremity at least 4 weeks prior,
* Severe spasticity in the upper extremity (Modified Ashworth Scale ≥3),
* Presence of dysphagia or aphasia,
* Presence of cardiac problems such as atrial fibrillation, atrial flutter, sick sinus syndrome, or atrioventricular block.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Evaluation (FM-UE) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  We will use the Fugl-Meyer Upper Motor Assessment score, which is the most sensitive for treatment outcomes in stroke patients presenting with unilateral paresis in the post-stroke period. It measures upper extremity use and impairment, measuring shoulder, elbow, forearm, wrist, finger, and reflex movements from proximal to distal, synergistic to extrinsic. The score ranges from 0 to 66 and consists of 33 items. 0-28 indicates severe motor impairment; 29-42 indicates moderate motor impairment; and 43-66 indicates mild motor impairment. Higher scores indicate better performance. The FM-UE consists of one component, each rated on a 3-point ordinal scale (0=not achieved, 1=partially contributed, 2=completely contributed). The minimum clinically meaningful change on the FM-UE for chronic stroke has been determined to be 4.25 to 7.25. Consistent with the literature, we define an improvement of at least 6 points or more as significant.
Box and Block Test (BBT) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  The Box and Block Test is a manual dexterity test used to assess upper extremity motor function. It primarily assesses gross motor function. It is calculated by the number of 2.5 cm3 blocks thrown from one side to the other in 1 minute. A box and block test kit has been prepared to meet international standards.

SECONDARY OUTCOMES:
Hand Grip Strength | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  Grip strength on the affected side will be measured with a Jamar Hydraulic Dynamometer. The measurement protocol will be explained and demonstrated to the participant by an experienced physiotherapist. The dynamometer grip size will be adjusted to the participant's hand size, and the participant will be asked to squeeze the dynamometer for a practice trial. Anti-gravity support will be provided to maintain the position if necessary. Grip strength measurements with the Jamar dynamometer have proven to be highly valid and reliable, and normative values have been published.
Stroke Impact Scale (SIS) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  The SIS 3.0 assesses function and quality of life based on subjective report in eight clinically important domains. It consists of two parts. The first part is the main scale of the IAS, which assesses multidimensional health-related quality of life (QOL) including strength, hand function, ADL/instrumental ADL, mobility, communication, emotion, memory/thinking, and social participation. It consists of 59 items, and each item is subjectively rated by stroke patients on a 5-point Likert-type scale according to their perceived difficulty with the item in the past week. The score for each domain is converted to a score out of 100, and the average scores for all domains are used to represent stroke patients' multidimensional health-related quality of life. The formula Domain Score = [(Average Item Score -1) / (5 -1) x 100] is used to convert each domain score. SIS 3.0 also includes assessment of post-stroke recovery using a 0-100 visual analog scale (0: no recovery, 100: complete recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Rüstem Mustafaoğlu, associate professor, Principal Investigator — Istanbul University-Cerrahpasa Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Fatih Aykut Çavdar, Study Chair — Marmara University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Yusuf Açıkgöz, Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; İpek Yeldan, Professor, Study Chair — Istanbul University-Cerrahpasa Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Belgin Erhan, Professor, Study Director — Istanbul Medeniyet University Faculty of Medicine, Department of International Medicine and Rehabilitation
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa Sağlık Bilimleri Fakültesi Büyükçekmece Yerleşkesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No